CLINICAL TRIAL: NCT00950950
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose Study to Evaluate the Effect of AMG 785 on Parameters of Bone Quality of the Forearm Using pQCT in Postmenopausal Women With Low Bone Mineral Density
Brief Title: A Study to Evaluate the Effect of Romosozumab (AMG 785) on Bone Quality of the Forearm in Postmenopausal Women With Low Bone Mass
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20090153
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-03

CONDITIONS: Osteopenia
Keywords: Amgen; Postmenopausal; Bone Density
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Participants were randomized to receive matching placebo administered by subcutaneous injection once every 4 weeks (Q4W) for 3 months.
  Interventions: Drug: Placebo
- Romosozumab (Experimental): Participants were randomized to receive 3 mg/kg romosozumab administered by subcutaneous injection once every 4 weeks (Q4W) for 3 months.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Administered by subcutaneous injection
  Other Names: AMG 785; EVENITY™
  Arms: Romosozumab
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of romosozumab on parameters of bone quality of the forearm using peripheral quantitative computed tomography (pQCT) following multiple subcutaneous dose administrations of romosozumab in postmenopausal women with low bone mass.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females between 55 to 80 years of age
* Postmenopausal females (based on medical history) defined as 12 continuous months of spontaneous amenorrhea

  * Women 60 years of age and older will be considered postmenopausal
  * Women 55-59 must have a serum follicle-stimulating hormone result > 40 mIU/mL and serum estradiol ≤ 20 pg/mL
* Low bone mineral density (BMD), defined as a BMD T-score between -1.0 and -2.5 at the lumbar spine (L1-L4) and/or femoral neck
* Weight ≤ 98 kg (216 lb) and/or height ≤ 196 cm (77 in)
* 25-hydroxyvitamin D ≥ 20 ng/mL at screening
* Willing and able to take ≥ 500 mg calcium and ≥ 400 IU (but ≤ 1,000 IU) vitamin D daily

Exclusion Criteria:

* Osteoporosis, defined as a BMD T-score ≤ -2.5 at the lumbar spine or femoral neck
* History of vertebral fracture, or fragility fracture of the wrist, humerus, hip or pelvis
* Diagnosed with any condition that will affect bone metabolism
* Subjects with fewer than 2 evaluable vertebrae; metal in forearms bilaterally that would not allow for at least one evaluable forearm
* Administration of the following medications within 6 months before study drug administration. This includes all routes of administration, for example intranasal and topical skin patches, unless otherwise noted:

  * Hormone replacement therapy [(eg, estrogen, estrogen-like compounds such as raloxifene). Infrequent use of estrogen vaginal creams (< 3 times per week) is allowed.]
  * Calcitonin
  * Parathyroid hormone (or any derivative)
  * Glucocorticosteroids (inhaled or topical corticosteroids administered more than 2 weeks before the enrollment date are allowed)
  * Anabolic steroids
  * Calcitriol, and available analogues
* Administration of daily, weekly, or monthly bisphosphonates (BP) unless meeting the following criteria:

  * < 2 weeks of BP use requires a 2-month washout period
  * 2 weeks to 3 months of BP use requires a 9-month washout period
  * 3 to 6 months of BP use requires a 1-year washout period
  * > 6 months of BP use requires a 3-year washout period;
* Greatly differing levels of physical activity or constant levels of intense physical exercise during the 6 months before study drug administration
* Known sensitivity to mammalian-derived drug preparations
* Known to be hepatitis B surface antigen, hepatitis C virus or human Immunodeficiency virus (HIV) positive or a known diagnosis of acquired immunodeficiency syndrome (AIDS)
* Any organic or psychiatric disorder, which, in the opinion of the investigator, poses a risk to subject safety and may prevent the subject from completing the study or interfere with the interpretation of the study results
* Unavailable for follow-up assessment or any concerns for subject's compliance with the protocol procedures
* Any other condition that might reduce the chance of obtaining data required by the protocol or that might compromise the ability to give truly informed consent
* History or evidence of a clinically significant disorder, condition or disease that, in the opinion of the Investigator or Amgen physician would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Clinically significant abnormality during the screening physical examination, electrocardiogram (ECG) or laboratory evaluation
* Participation in another clinical study within 4 weeks of screening or within 5 times the half-life of the investigational agent in the other clinical study, if known
* Has donated or lost 400 mL or more of blood or plasma within 8 weeks of study drug administration
* Previous AMG 785 exposure

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08-18 (Actual); Primary Completion 2010-08-19 (Actual); Study Completion 2010-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: Participants were equally randomized to receive romosozumab or placebo.
Period: Overall Study
Arm/Group | Placebo | Romosozumab
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romosozumab | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (5.6) | 65.6 (7.2) | 63.9 (6.5)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 9 | 6 | 15
  65 - 74 years | 3 | 4 | 7
  ≥ 75 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 12 | 24
Polar Moment of Inertia [Median (Full Range); unit: mm⁴] — The polar moment of inertia is a geometric measurement used to predict bone quality, specifically the ability to resist torsion (twisting), and is highly correlated with fracture load at the distal radius. The polar cross-sectional moment of inertia was assessed using peripheral quantitative computed tomography (pQCT), a 3-dimensional imaging technology which can be used for volumetric analysis of appendicular skeletal sites such as the arms and the legs. The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate.
  mm⁴ | 1545.14 [932.79 to 2045.53] | 1496.50 [1162.51 to 2059.27] | 1501.96 [932.79 to 2059.27]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Polar Cross-sectional Moment of Inertia at the Distal Radius
Description: The polar moment of inertia is a geometric measurement used to predict bone quality, specifically the ability to resist torsion (twisting), and is highly correlated with fracture load at the distal radius. The polar cross-sectional moment of inertia was assessed using peripheral quantitative computed tomography (pQCT), a 3-dimensional imaging technology which can be used for volumetric analysis of appendicular skeletal sites such as the arms and the legs. The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -1.16 (1.40) | 0.16 (0.95)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -1.03 (1.00) | -1.03 (1.19)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -2.28 (1.21) | 1.45 (1.03)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -1.93 (1.22) | 0.87 (0.89)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -1.66 (1.22) | -0.08 (1.12)

2. Secondary Outcome: Percent Change From Baseline in Total Bone Area at the Distal Radius
Description: Total bone area was assessed using peripheral quantitative computed tomography (pQCT), a 3-dimensional imaging technology which can be used for volumetric analysis of appendicular skeletal sites such as the arms and the legs. The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.07 (0.56) | -0.21 (0.40)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.08 (0.48) | -0.13 (0.56)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -0.79 (0.49) | 0.38 (0.61)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | 0.05 (0.43) | 0.87 (0.66)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -0.23 (0.46) | -0.04 (0.70)

3. Secondary Outcome: Percent Change From Baseline in Total Bone Mineral Content at the Distal Radius
Description: Total bone mineral content was assessed using peripheral quantitative computed tomography (pQCT). The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.39 (0.40) | -0.27 (0.41)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.33 (0.37) | -0.49 (0.27)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -0.86 (0.47) | -0.51 (0.36)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -0.66 (0.36) | -0.43 (0.37)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -1.34 (0.30) | -1.09 (0.36)

4. Secondary Outcome: Percent Change From Baseline in Total Bone Mineral Density at the Distal Radius
Description: Total bone mineral density was assessed using peripheral quantitative computed tomography (pQCT). The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.30 (0.48) | -0.06 (0.30)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.24 (0.38) | -0.34 (0.44)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -0.07 (0.19) | -0.86 (0.53)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -0.69 (0.48) | -1.26 (0.53)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -0.10 (0.42) | -1.02 (0.55)

5. Secondary Outcome: Percent Change From Baseline in Cortical Bone Area at the Distal Radius
Description: Cortical bone area was assessed using peripheral quantitative computed tomography (pQCT). The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.27 (0.58) | 0.06 (0.63)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.05 (0.54) | -0.53 (0.64)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -1.39 (0.77) | 0.69 (0.67)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -1.41 (0.81) | 0.28 (0.63)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -1.59 (0.58) | -0.50 (0.74)

6. Secondary Outcome: Percent Change From Baseline in Cortical Bone Mineral Content at the Distal Radius
Description: Cortical bone mineral content was assessed using peripheral quantitative computed tomography (pQCT). The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.33 (0.57) | 0.07 (0.46)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.29 (0.52) | -0.86 (0.45)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -1.08 (0.66) | -0.07 (0.66)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -1.45 (0.82) | -0.66 (0.57)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -1.69 (0.55) | -1.29 (0.67)

7. Secondary Outcome: Percent Change From Baseline in Cortical Bone Mineral Density at the Distal Radius
Description: Cortical bone mineral density was assessed using peripheral quantitative computed tomography (pQCT). The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.06 (0.10) | 0.02 (0.21)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.24 (0.21) | -0.32 (0.28)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 0.32 (0.24) | -0.76 (0.23)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -0.04 (0.23) | -0.92 (0.40)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -0.10 (0.23) | -0.79 (0.31)

8. Secondary Outcome: Percent Change From Baseline in Endocortical Circumference at the Distal Radius
Description: Endocortical circumference was derived from pQCT measurements based on applying a circular ring model to the cortical shell. The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | 0.20 (0.74) | -0.19 (0.50)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.23 (0.73) | 0.26 (0.67)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -0.03 (0.39) | -0.07 (0.72)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | 0.77 (0.80) | 0.89 (0.66)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | 0.85 (0.66) | 0.49 (0.84)

9. Secondary Outcome: Percent Change From Baseline in Periosteal Circumference at the Distal Radius
Description: Periosteal circumference was derived from pQCT measurements based on applying a circular ring model to the cortical shell. The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.04 (0.28) | -0.11 (0.20)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.04 (0.24) | -0.07 (0.28)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -0.40 (0.25) | 0.19 (0.31)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | 0.02 (0.22) | 0.43 (0.33)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -0.12 (0.23) | -0.02 (0.35)

10. Secondary Outcome: Percent Change From Baseline in Cortical Thickness at the Distal Radius
Description: Cortical thickness was derived from pQCT measurements based on applying a circular ring model to the cortical shell. The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.29 (0.82) | 0.22 (0.77)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | 0.09 (0.79) | -0.56 (0.85)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -1.14 (0.72) | 0.64 (0.99)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -1.69 (1.14) | -0.31 (0.80)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -1.82 (0.78) | -0.62 (1.09)

11. Secondary Outcome: Percent Change From Baseline in Polar Section Modulus at the Distal Radius
Description: Polar section modulus is a measurement of bone strength and was derived from pQCT measurements. The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | 0.18 (0.78) | 0.02 (0.78)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.11 (1.08) | -0.46 (1.05)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -2.14 (1.40) | 0.93 (1.22)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -2.31 (1.55) | 1.76 (1.32)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -1.67 (1.14) | -1.05 (1.20)

12. Secondary Outcome: Percent Change From Baseline in Polar Strength Strain Index at the Distal Radius
Description: The polar strength strain index is a measurement of bone strength and was derived from pQCT measurements. The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -1.85 (0.81) | -0.78 (0.51)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -1.32 (0.75) | -1.47 (1.21)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 0.36 (0.99) | -1.91 (1.49)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -0.71 (0.95) | -1.57 (0.94)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -0.41 (0.98) | -1.25 (0.78)

13. Secondary Outcome: Percent Change From Baseline in Axial Moment of Inertia at the Distal Radius
Description: Axial moment of inertia is an indicator of the ability of bone to resist bending, and was derived from pQCT measurements based on a circular ring model. The distal slice was acquired at 20% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.22 (0.91) | -0.23 (0.73)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -0.19 (0.74) | -0.49 (0.88)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -1.90 (1.09) | 0.94 (0.83)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -0.90 (0.65) | 1.41 (1.04)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -1.25 (0.75) | -0.28 (0.98)

14. Secondary Outcome: Percent Change From Baseline in Total Bone Area at the Ultradistal Radius
Description: Total bone area was assessed using peripheral quantitative computed tomography (pQCT), a 3-dimensional imaging technology which can be used for volumetric analysis of appendicular skeletal sites such as the arms and the legs. The ultradistal slice was acquired at 4% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -2.30 (3.64) | -0.72 (2.35)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -5.11 (2.44) | -0.01 (3.66)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -0.27 (2.37) | 7.35 (3.21)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -0.43 (2.46) | 3.27 (2.96)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | 1.90 (2.50) | 0.91 (3.32)

15. Secondary Outcome: Percent Change From Baseline in Total Bone Mineral Content at the Ultradistal Radius
Description: Total bone mineral content was assessed using peripheral quantitative computed tomography (pQCT). The ultradistal slice was acquired at 4% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | 0.63 (0.43) | -0.30 (0.70)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | 0.13 (0.53) | -0.09 (0.63)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 0.63 (0.56) | 1.16 (0.39)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | 0.46 (0.56) | -0.14 (0.46)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | 0.15 (0.59) | -0.64 (0.97)

16. Secondary Outcome: Percent Change From Baseline in Total Bone Mineral Density at the Ultradistal Radius
Description: Total bone mineral density was assessed using peripheral quantitative computed tomography (pQCT). The ultradistal slice was acquired at 4% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | 4.45 (4.42) | 0.91 (1.97)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | 6.22 (3.19) | 1.19 (2.98)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 1.52 (2.64) | -4.95 (2.33)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | 1.43 (2.35) | -2.53 (2.38)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -1.14 (2.72) | -0.81 (2.59)

17. Secondary Outcome: Percent Change From Baseline in Trabecular Bone Area at the Ultradistal Radius
Description: Trabecular bone area was assessed using peripheral quantitative computed tomography (pQCT). The ultradistal slice was acquired at 4% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -3.54 (5.68) | -0.64 (3.59)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -8.06 (3.86) | 0.43 (6.21)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -0.55 (3.82) | 12.00 (5.84)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -1.86 (4.01) | 5.60 (5.22)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | 2.84 (4.18) | 1.57 (5.20)

18. Secondary Outcome: Percent Change From Baseline in Trabecular Bone Mineral Content at the Ultradistal Radius
Description: Trabecular bone mineral content was assessed using peripheral quantitative computed tomography (pQCT). The ultradistal slice was acquired at 4% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -3.26 (7.35) | -0.52 (4.78)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -9.52 (4.68) | 0.02 (7.61)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 1.02 (5.51) | 14.64 (7.06)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -0.70 (6.15) | 5.68 (6.54)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | 5.12 (5.55) | 1.74 (6.71)

19. Secondary Outcome: Percent Change From Baseline in Trabecular Bone Mineral Density at the Ultradistal Radius
Description: Trabecular bone mineral density was assessed using peripheral quantitative computed tomography (pQCT). The ultradistal slice was acquired at 4% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | -0.78 (1.88) | -0.34 (1.33)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -1.98 (1.16) | -1.30 (1.59)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 0.98 (1.64) | 2.00 (0.88)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | 0.53 (1.92) | -0.49 (1.19)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | 1.74 (1.47) | -0.51 (1.64)

20. Secondary Outcome: Percent Change From Baseline in Polar Strength Strain Index at the Ultradistal Radius
Description: The polar strength strain index is a measurement of bone strength and was derived from pQCT measurements. The ultradistal slice was acquired at 4% of the length of the ulna proximal to the radial endplate. Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 10 | 11
  Day 29 | 2.69 (2.36) | -0.14 (1.00)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | 2.28 (1.47) | 1.28 (2.06)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 1.08 (1.71) | -0.90 (2.30)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -0.87 (1.29) | -0.89 (1.95)
  Day 169: number analyzed (Participants) | 11 | 10
  Day 169 | -0.25 (1.61) | -1.51 (1.86)

21. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the One-third Radius
Description: Bone mineral density was assessed using dual energy x-ray absorptiometry (DXA). Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 11 | 12
  Day 29 | 1.715 (0.808) | 1.210 (0.814)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | 0.832 (1.155) | -0.694 (0.827)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 0.790 (1.117) | -1.941 (0.986)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -0.118 (1.405) | -0.439 (1.346)
  Day 169: number analyzed (Participants) | 11 | 11
  Day 169 | 1.866 (0.905) | -0.328 (0.702)

22. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Total Wrist
Description: Bone mineral density was assessed using dual energy x-ray absorptiometry (DXA). Scans were analyzed by a central reader.
Time Frame: Baseline and days 29, 57, 85, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 29: number analyzed (Participants) | 11 | 12
  Day 29 | 1.829 (0.617) | -0.555 (0.428)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | 0.940 (1.081) | -1.651 (0.574)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 0.233 (0.996) | -1.690 (0.733)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | 0.001 (1.081) | -0.369 (0.765)
  Day 169: number analyzed (Participants) | 11 | 11
  Day 169 | 0.357 (1.237) | -0.649 (0.522)

23. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density at the Total Lumbar Spine
Description: Bone mineral density was assessed using dual energy x-ray absorptiometry (DXA). Scans were analyzed by a central reader.
Time Frame: Baseline and days 85 and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 0.345 (1.224) | 4.786 (0.846)
  Day 169: number analyzed (Participants) | 11 | 11
  Day 169 | 0.149 (0.905) | 7.876 (1.351)

24. Secondary Outcome: Percent Change From Baseline in Serum Procollagen Type 1 N-terminal Propeptide (P1NP)
Time Frame: Baseline and days 4, 15, 29, 57, 62, 71, 85, 99, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 4: number analyzed (Participants) | 11 | 12
  Day 4 | -4.40 (6.13) | 36.37 (10.02)
  Day 15: number analyzed (Participants) | 11 | 12
  Day 15 | 3.46 (5.64) | 146.39 (20.00)
  Day 29: number analyzed (Participants) | 11 | 12
  Day 29 | -0.33 (3.44) | 101.85 (19.97)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | -6.93 (4.52) | 74.77 (10.91)
  Day 62: number analyzed (Participants) | 11 | 11
  Day 62 | 0.27 (9.20) | 92.22 (14.71)
  Day 71: number analyzed (Participants) | 11 | 11
  Day 71 | 19.61 (16.22) | 106.91 (14.08)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | 23.83 (17.11) | 67.85 (19.11)
  Day 99: number analyzed (Participants) | 11 | 11
  Day 99 | 10.94 (15.57) | 17.07 (11.79)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | 5.49 (10.26) | 12.56 (8.57)
  Day 169: number analyzed (Participants) | 11 | 11
  Day 169 | 20.85 (10.44) | 33.80 (13.64)

25. Secondary Outcome: Percent Change From Baseline in Serum C-Telopeptide (sCTX)
Time Frame: Baseline and days 4, 15, 29, 57, 62, 71, 85, 99, 127, and 169
Population: Treated participants with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab
Number analyzed (Participants) | 12 | 12
percent change
  Day 4: number analyzed (Participants) | 11 | 12
  Day 4 | 6.62 (4.33) | -23.77 (7.78)
  Day 15: number analyzed (Participants) | 11 | 12
  Day 15 | -2.29 (5.15) | -33.10 (8.85)
  Day 29: number analyzed (Participants) | 11 | 12
  Day 29 | -3.19 (8.83) | -21.42 (13.98)
  Day 57: number analyzed (Participants) | 11 | 12
  Day 57 | 7.87 (6.49) | 7.26 (16.28)
  Day 62: number analyzed (Participants) | 11 | 11
  Day 62 | 8.69 (5.78) | -12.67 (15.15)
  Day 71: number analyzed (Participants) | 11 | 11
  Day 71 | 5.60 (5.59) | -14.72 (13.84)
  Day 85: number analyzed (Participants) | 11 | 11
  Day 85 | -3.00 (7.94) | 4.85 (19.28)
  Day 99: number analyzed (Participants) | 11 | 11
  Day 99 | -9.14 (8.17) | 14.29 (23.73)
  Day 127: number analyzed (Participants) | 11 | 11
  Day 127 | -10.00 (8.91) | 6.32 (16.60)
  Day 169: number analyzed (Participants) | 11 | 11
  Day 169 | -3.61 (8.95) | 16.06 (20.53)

26. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of Romosozumab
Description: Serum concentrations of romosozumab were measured by a validated enzyme-linked immunosorbent assay. The lower limit of quantification (LLOQ) was 50 ng/mL.
Time Frame: First Dose: Day 1 (predose) and on days 4, 15, and 29 (predose). Last Dose: Days 57 (predose), 62, 71, 85, 99, 127, and 169
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be calculated
Measure: Median (Full Range); unit: days
Arm/Group | Romosozumab
Number analyzed (Participants) | 12
days
  First dose | 3.0 [3.0 to 3.0]
  Last dose: number analyzed (Participants) | 11
  Last dose | 5.0 [5.0 to 14]

27. Secondary Outcome: Maximum Serum Concentration (Cmax) of Romosozumab
Description: as for outcome 26
Time Frame: as for outcome 26
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be calculated
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Romosozumab
Number analyzed (Participants) | 12
μg/mL
  First dose | 26.8 (6.4)
  Last dose: number analyzed (Participants) | 11
  Last dose | 32.3 (9.6)

28. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Tau (AUC0-28)
Description: Serum concentrations of romosozumab were measured by a validated enzyme-linked immunosorbent assay. The lower limit of quantification (LLOQ) was 50 ng/mL.
  The area under the serum drug concentration-time curve from time zero to tau (tau = 28 days) (AUC0-28) was calculated by the linear trapezoidal method.
Time Frame: as for outcome 26
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be calculated
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Romosozumab
Number analyzed (Participants) | 12
μg*day/mL
  First dose | 422 (75)
  Last dose: number analyzed (Participants) | 11
  Last dose | 501 (179)

29. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUCinf)
Description: as for outcome 26
Time Frame: Last Dose: Days 57 (predose), 62, 71, 85, 99, 127, and 169
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be calculated
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Romosozumab
Number analyzed (Participants) | 11
μg*day/mL | 590 (240)

30. Secondary Outcome: Apparent Clearance (CL/F) of Romosozumab
Description: as for outcome 26
Time Frame: Last Dose: Days 57 (predose), 62, 71, 85, 99, 127, and 169
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be calculated
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Romosozumab
Number analyzed (Participants) | 11
mL/day/kg | 5.82 (2.12)

31. Secondary Outcome: Terminal Half-life (t1/2,z) of Romosozumab
Description: as for outcome 26
Time Frame: Last Dose: Days 57 (predose), 62, 71, 85, 99, 127, and 169
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be calculated
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Romosozumab
Number analyzed (Participants) | 11
days | 6.82 (0.92)

32. Secondary Outcome: Accumulation Ratio
Description: Accumulation ratio was calculated as the ratio of AUC0-28 after the last dose to AUC0-28 after the first dose.
Time Frame: as for outcome 26
Population: All participants who received romosozumab and for whom the pharmacokinetic parameter could be calculated
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Romosozumab
Number analyzed (Participants) | 11
ratio | 1.15 (0.27)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Placebo: Participants received matching placebo administered by subcutaneous injection once every 4 weeks (Q4W) for 3 months.
- Romosozumab: Participants received 3 mg/kg romosozumab administered by subcutaneous injection once every 4 weeks (Q4W) for 3 months.
Arm/Group | Placebo | Romosozumab
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/12
Other Adverse Events (participants affected / at risk) | 10/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Romosozumab (N=12)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Romosozumab (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Injection site discomfort (General disorders) | 1 | 0
Injection site reaction (General disorders) | 2 | 1
Injection site swelling (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Thrombophlebitis superficial (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.